CLINICAL TRIAL: NCT00469456
Title: A Randomized, Double-Blind, Placebo-Controlled Evaluation of the Efficacy of Memantine on Functional Communication in Patients With Alzheimer's Disease (AD)
Brief Title: Effect of Memantine on Functional Communication in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Stephen Graham, PhD, Sr. Director, Forest Research Institute, a division of Forest Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEM-MD-71
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Results first posted 2009-12-07 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Alzheimer's Disease
Keywords: memantine; Alzheimer's Disease; communication
MeSH Terms: conditions — Alzheimer Disease; Communication | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Active Comparator): Memantine 20mg (10mg twice daily) oral administration for 12 weeks
  Interventions: Drug: Memantine
- 2 (Placebo Comparator): Placebo oral administration twice daily for 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Memantine — Memantine 20mg (10mg twice daily) oral administration for 12 weeks
  Other Names: Namenda®
  Arms: 1
Drug: placebo — Placebo oral administration twice daily for 12 weeks
  Arms: 2

SUMMARY:
The objective of this study is to evaluate the effect of memantine versus placebo on functional communication in patients with Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, 50 years or older, native English speakers, meeting National Institute of Neurological and Communicative Disorders and Stroke--Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for probable AD with a Mini Mental State Examination (MMSE) score of 10 to 19 at Screening and Baseline

Exclusion Criteria:

* Current Diagnostic and Statistical Manual of Mental Disorders--Fourth Edition (DSM-IV) Axis I disorder other than AD
* Previous imaging results not consistent with the diagnosis of AD
* Modified Hachinski Ischemia Score greater than 4
* Evidence of other neurologic disorders
* Clinically significant systemic disease
* A known or suspected history of alcohol or drug abuse in the past 5 years
* Taking excluded medication
* Previous treatment with commercial memantine

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F C Potocnik, Principal Investigator
Locations (23):
- Australia (14):
  - Forest Investigative Site, East Gosford, New South Wales
  - Forest Investigative Site, Hornsby, New South Wales
  - Forest Investigative Site, Kogarah, New South Wales
  - Forest Investigative Site, Newcastle, New South Wales
  - Forest Investigative Site, Randwick, New South Wales
  - Forest Investigative Site, Chermside, Queensland
  - Forest Investigative Site, Toowoomba, Queensland
  - Forest Investigative Site, Adelaide, South Australia
  - Forest Investigative Site, Woodville, South Australia
  - Forest Investigative Site, Box Hill, Victoria
  - Forest Investigative Site, Frankston, Victoria
  - Forest Investigative Site, Heidelberg West, Victoria
  - Forest Investigative Site, Kew, Victoria
  - Forest Investigative Site, Perth, Western Australia
- New Zealand (3):
  - Forest Investigative Site, Christchurch
  - Forest Investigative Site, North Shore
  - Forest Investigative Site, Timaru
- South Africa (6):
  - Forest Investigative Site, George, E. Cape
  - Forest Investigative Site, Port Elizabeth, E. Cape
  - Forest Investigative Site, Johannesburg, Gauteng
  - Forest Investigative Site, Pretoria, Gauteng
  - Forest Investigative Site, Durban, KZ-Natal
  - Forest Investigative Site, Cape Town, W. Cape

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from May 24, 2007 to July 29, 2008 at 25 centers in three countries [14 in Australia, 3 in New Zealand, 8 in South Africa].
Pre-assignment Details: Study consisted of up to 2 weeks single-blind placebo treatment followed by 12 weeks double-blind treatment. At end of single-blind placebo treatment, patients (pts) meeting entry criteria were randomized (1:1) to 1 of 2 double-blind treatment groups receiving memantine or placebo. Pts not meeting inclusion/exclusion criteria were not randomized.
Groups:
- Placebo: Matching placebo, oral administration, twice daily for 12 weeks
- Memantine: Memantine 20mg (10mg twice daily), oral administration for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Memantine
Started | 129 (Safety Population defined as all patients who took at least one dose of double-blind study drug) | 135 (Safety Population defined as all patients who took at least one dose of double-blind study drug.)
Completed | 120 | 131
Not Completed | 9 | 4
Not completed — Adverse Event | 4 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Memantine | Total
Number analyzed (Participants) | 129 | 135 | 264
Age, Customized [Number; unit: participants]
  <=64 years | 19 | 13 | 32
  65-74 years | 33 | 51 | 84
  75-84 years | 59 | 56 | 115
  >=85 years | 18 | 15 | 33
Age Continuous [Mean (Standard Deviation); unit: years] | 75.1 (8.68) | 74.8 (8.05) | 74.9 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants] — One patient was randomized but did not receive study drug.
  Participants
    Female | 74 | 80 | 154
    Male | 55 | 55 | 110
Region of Enrollment [Number; unit: participants]
  Australia | 55 | 55 | 110
  South Africa | 58 | 62 | 120
  New Zealand | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Functional Linguistic Communication Inventory (FLCI) at Week 12
Description: FLCI is a standardized & validated instrument for evaluating functional communication in pts with moderate-to-severe Alzheimer's that can be used to obtain Baseline information & to track patients' capabilities thereafter. The FLCI evaluates 10 areas: greeting and naming, answering questions, writing, sign comprehension, object-to-picture matching, word reading and comprehension, following commands, pantomime, gesture, and conversation. The FLCI total score ranges from 0 to 87, a higher score denotes better functional communication, and takes approximately 30 minutes to complete.
Time Frame: Baseline to Week 12
Population: Primary efficacy analysis was based on the Intent-to-Treat (ITT) Population. The ITT Population will consist of all patients in the Safety Population who had at least one post-Baseline assessment of the primary efficacy parameter, FLCI. The last-observation-carried-forward approach was used to impute missing post-Baseline values.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 124 | 133
Units on a scale | -0.6 (0.59) | 0.7 (0.57)
Statistical Analysis 1: Comparison: Placebo vs Memantine; The primary efficacy parameter was change from Baseline to Week 12 in FLCI total score. Missing FLCI total scores at Week 12 were imputed using the last-observation-carried-forward (LOCF) approach; Test type: Superiority or Other; p = 0.070, ANCOVA; Mean Difference (Final Values) = 1.3, 95% CI [-0.1 to 2.8]

2. Secondary Outcome: Change From Baseline in American Speech-Language-Hearing Association Functional Assessment of Communication Skills for Adults (ASHA FACS) [Total Score of Social Communication and Communication of Basic Needs Subscores] at Week 12
Description: The ASHA FACS assesses & measures functional communication skills of adults with speech, language, & cognitive communication disorders. The measure, which comprises 43 items and takes approximately 20 minutes to complete, assesses functional communication in four areas: social communication; communication of basic needs; reading, writing, and number concepts; and daily planning. Total score of subdomains [Social Communication and Communication of Basic Needs] ranges from 0-196. A higher score denotes better communication.
Time Frame: Baseline to Week 12
Population: The secondary efficacy analysis was based on the ITT Population. The last-observation-carried-forward approach was used to impute missing post-Baseline values.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 124 | 133
Units on a scale | -5.3 (2.06) | 0.5 (1.99)
Statistical Analysis 1: Comparison: Placebo vs Memantine; The secondary efficacy parameter was change from Baseline at Week 12 in the total score of the Social Communication subscale and Communication of Basic Needs subscale of the ASHA FACS. Missing scores at week 12 were imputed using the last-observation-carried-forward (LOCF) approach; Test type: Superiority or Other; p = 0.022, ANCOVA; Mean Difference (Final Values) = 5.9, 95% CI [0.9 to 10.9]

ADVERSE EVENTS:
Time Frame: Occurring on or after the date of the first dose of double-blind study medication and within 30 days of the date of last dose of double-blind study medication.
Arm/Group | Placebo | Memantine
Serious Adverse Events (participants affected / at risk) | 13/129 | 4/135
Other Adverse Events (participants affected / at risk) | 2/129 | 7/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=129) | Memantine (N=135)
Syncope (Nervous system disorders) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 1
Atrioventricular Block First Degree (Cardiac disorders) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cerebellar Infarction (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointeritis Yersinia (Infections and infestations) | 1 | 0
Hiatus Hernia (Gastrointestinal disorders) | 1 | 0
Pneumonia Aspiration (Infections and infestations) | 0 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Vestibular Disorder (Ear and labyrinth disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=129) | Memantine (N=135)
Dizziness (Nervous system disorders) | 2 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 90 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential info. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in pub. On sponsor's request, PI shall delay submission for any pub while sponsor files patent apps. If trial is multi-center, PI agrees that first publication shall be a multi-center pub.